CLINICAL TRIAL: NCT05822414
Title: Erector Spinae Plane Block Vs. Superior Trunk Block for Postoperative Pain Control After Arthroscopic Shoulder Surgery: a Randomized Controlled Trial
Brief Title: ESP Vs STB for Pain and Diaphragm Function for Shoulder Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 202301211RINB
Record Dates: First submitted 2023-04-10; First posted 2023-04-20 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Rotator Cuff Injuries
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Erector Spinae Plane Block group (Experimental)
  Interventions: Procedure: Erector spinae plane block
- Superior Trunk Block group (Active Comparator)
  Interventions: Procedure: Erector spinae plane block

INTERVENTIONS:
Procedure: Erector spinae plane block — Erector spinae plane block will be injected at the second thoracic vertebral level for patient undergoing rotator cuff repair surgery

SUMMARY:
To compare the efficacy of pain control, shoulder function recovery, and degree of diaphragm palsy between erector spinae plane block at T2 level and superior trunk block after arthroscopic shoulder surgery

DETAILED DESCRIPTION:
Arthroscopic shoulder surgery can cause a substantial degree of postoperative pain that interferes with postoperative recovery. Adequate perioperative pain control can not only decrease duration of hospital length of stay and prevent unnecessary re-admission, but also facilitate postoperative rehabilitation and improve overall quality of life.

According to the 2019 PROSPECT guideline for rotator cuff repair surgery: systematic review and procedure-specific postoperative pain management recommendations, published on Anesthesia, postoperative pain can be controlled by systemic analgesics such as paracetamol and NSAIDS, regional analgesia, and opioids as rescue analgesia.

The current nerve block of choice is the interscalene brachial plexus block. It can provide adequate pain control, but is associated with several drawbacks including neurological injuries from direct nerve contact and pneumothorax, with the potential for phrenic nerve blockade and hemidiaphragmatic paresis raising the most concern. The superior trunk block, which is performed at where the C5 and C6 roots converge to form the superior trunk, was therefore developed, as it is located further away from the phrenic nerve. However, there are still considerable risks of phrenic nerve blockade, as well as nerve injury from direct contact and upper limb motor blockade.

The erector spinae plane block, first described by Forero et al. in 2016, involves the injection of local anaesthetic deep to the erector spinae muscles and has been widely studied for analgesia in thoracic surgery. It is a paraspinal fascial plane block and is assumed to share the same mechanism at different vertebral levels, including cervical and lumbar, to provide analgesia for a variety of different surgeries, including spine and breast surgeries. In recent years, erector spinae plane block performed at T2 level has also been employed for chronic shoulder pain and arthroscopic shoulder surgery perioperative pain management. Significant better perioperative pain control was achieved when compared with sham block using normal saline by Cftci et al. in 2021 and non inferior pain control was achieved when compared with peri-articular injection of local anesthetics by Shanthanna et al in 2022.

To date, there is no head to head trial comparing the effect of the established block of choice, interscalene brachial plexus block or superior trunk block, to the more novel T2 erector spinae plane block. We therefore designed this study to compare the use of superior trunk block and T2 erector spinae plane block in arthroscopic shoulder surgery with respect to their respective analgesic efficacy and undesired side effect of hemidiaphragm palsy. Primary outcomes of the study are postoperative pain score evaluated by the 100mm-visual analogue scale and morphine consumption, and diaphragm excursion assessed with ultrasonography, while the secondary outcomes include patient reported outcomes assessed by Quality of Recovery-15 (QOR-15) and Shoulder Pain and Disability Index (SPADI)

ELIGIBILITY:
Inclusion Criteria:

* patients receiving arthroscopic shoulder surgery

Exclusion Criteria:

* patients with age <18 and >85
* pregnancy
* patients with severe organ failure: respiratory failure (FEV1 (Forced expiratory volume) /FVC (forced vital capacity)<70% and FEV1< 50%), heart failure (NYHA class III, IV), renal failure (eGFR<60ml/min/1.73m^2)
* patients diagnosed with chronic obstructive lung disease
* patients with arrhythmia
* patients with ongoing infection
* patients with chronic opioid use or substance abuse history
* patients with coagulopathy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-05-04 (Actual); Primary Completion 2024-12-11 (Actual); Study Completion 2024-12-11 (Actual)

PRIMARY OUTCOMES:
Assessment of postoperative pain severity | one hour and 24-hour after surgery
  Postoperative pain severity evaluated by 100mm-visual analogue scale (0-100; 0 means no pain at all and 100 means the worst pain intensity)
Assessment of diaphragm movement after block performance | before surgery and one hour after surgery
  Diaphragm movement evaluated by ultrasonography

SECONDARY OUTCOMES:
Assessment of postoperative quality of recovery | before surgery and 24 hours after surgery
  Postoperative quality of recovery evaluated by quality of recovery 15 (QoR-15)

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Yu Wu, MD, Study Chair — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kang R, Jeong JS, Chin KJ, Yoo JC, Lee JH, Choi SJ, Gwak MS, Hahm TS, Ko JS. Superior Trunk Block Provides Noninferior Analgesia Compared with Interscalene Brachial Plexus Block in Arthroscopic Shoulder Surgery. Anesthesiology. 2019 Dec;131(6):1316-1326. doi: 10.1097/ALN.0000000000002919. PMID 31490292
- [Background] Hussain N, Goldar G, Ragina N, Banfield L, Laffey JG, Abdallah FW. Suprascapular and Interscalene Nerve Block for Shoulder Surgery: A Systematic Review and Meta-analysis. Anesthesiology. 2017 Dec;127(6):998-1013. doi: 10.1097/ALN.0000000000001894. PMID 28968280
- [Background] Forero M, Rajarathinam M, Adhikary SD, Chin KJ. Erector spinae plane block for the management of chronic shoulder pain: a case report. Can J Anaesth. 2018 Mar;65(3):288-293. doi: 10.1007/s12630-017-1010-1. Epub 2017 Nov 13. PMID 29134518
- [Background] Shanthanna H, Czuczman M, Moisiuk P, O'Hare T, Khan M, Forero M, Davis K, Moro J, Vanniyasingam T, Foster G, Thabane L, Alolabi B. Erector spinae plane block vs. peri-articular injection for pain control after arthroscopic shoulder surgery: a randomised controlled trial. Anaesthesia. 2022 Mar;77(3):301-310. doi: 10.1111/anae.15625. Epub 2021 Dec 3. PMID 34861745
- [Background] Ciftci B, Ekinci M, Golboyu BE, Kapukaya F, Atalay YO, Kuyucu E, Demiraran Y. High Thoracic Erector Spinae Plane Block for Arthroscopic Shoulder Surgery: A Randomized Prospective Double-Blind Study. Pain Med. 2021 Apr 20;22(4):776-783. doi: 10.1093/pm/pnaa359. PMID 33155041
- [Background] Padua R, de Girolamo L, Grassi A, Cucchi D. Choosing patient-reported outcome measures for shoulder pathology. EFORT Open Rev. 2021 Sep 14;6(9):779-787. doi: 10.1302/2058-5241.6.200109. eCollection 2021 Sep. PMID 34667649
- [Background] Stark PA, Myles PS, Burke JA. Development and psychometric evaluation of a postoperative quality of recovery score: the QoR-15. Anesthesiology. 2013 Jun;118(6):1332-40. doi: 10.1097/ALN.0b013e318289b84b. PMID 23411725